CLINICAL TRIAL: NCT01849406
Title: A Randomized Crossover Trial of the Effect of Nasal Steroids in Snoring Intensity
Brief Title: Effect of Nasal Steroids in Snoring Intensity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ioannis Koutsourelakis (Other)
Responsible Party: Sponsor-Investigator, Ioannis Koutsourelakis, MD, PhD, University of Athens
Organization: University of Athens (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NASTER
Record Dates: First submitted 2013-04-14; First posted 2013-05-08 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring | interventions — Budesonide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal spray Budesonide (Active Comparator): one week therapy of nasal budesonide (twice per day)
  Interventions: Drug: nasal spray Budesonide
- Nasal spray Normal Saline (Placebo Comparator): one week therapy of nasal normal saline (twice per day)
  Interventions: Drug: Nasal spray Normal Saline

INTERVENTIONS:
Drug: nasal spray Budesonide — one week therapy of nasal budesonide twice per day
  Other Names: budesonide
  Arms: Nasal spray Budesonide
Drug: Nasal spray Normal Saline — one week therapy of nasal normal saline twice per day
  Other Names: Normal saline
  Arms: Nasal spray Normal Saline

SUMMARY:
It is anecdotally well known that patients snore more when their nose is blocked. However, the therapeutic effect of improving nasal airway patency on snoring indices remains a point of conjecture. Indeed, Braver et al examined the effect of a nasal vasoconstrictor and failed to show any improvement in the number of snores after its application, although apnoea-hypopnoea index (AHI)seemed to decrease. Furthermore, Hoffstein et al documented that dilation of the anterior nares in patients without nasal pathology has a relatively weak effect on snoring, and routine use of nasal dilating appliances was not recommended for the treatment of snoring. In contrast to the aforementioned studies, intranasal corticosteroids have been shown to improve sleepiness and reduce AHI in patients with obstructive sleep apnea (OSA) implying that there might be an equivalent result for the use of nasal steroids on snoring indices.

Additionally, the present authors have demonstrated a strong correlation between apnoea-hypopnoea index and oral/oro-nasal breathing epochs in patients with OSA and normal nasal resistance and that nasal surgery is effective only in OSA patients who preoperatively have decreased nasal breathing epochs.

It is plausible thus to suggest that snoring severity, in equivalence to OSA severity, might be associated to oral/oro-nasal breathing epochs and that improving nasal patency by nasal steroids might also increase nasal breathing epochs and lead to decreased snoring indices in patients who had decreased nasal breathing before the administration of nasal steroids.

Patients will be randomized in two groups: the patients of the first group will undergo a one week therapy of nasal budesonide, then two weeks of washout period, and thereafter one week of nasal normal saline. The patients of the second group will undergo a one week therapy of nasal normal saline, then two weeks of washout period, and thereafter one week of nasal budesonide. Before and after each treatment regimen patients will undergo an assessment, which will consist of anterior rhinomanometry and polysomnography with concomitant measurement of snoring indices and breathing route pattern.

The investigators hypothesize that the application for one week of nasal budesonide has a beneficial effect on snoring indices in patients who present before the application decreased proportion of nasal breathing epochs and in whom nasal budesonide succeeded in increasing nasal breathing epochs.

DETAILED DESCRIPTION:
Snoring intensity would be measured using a calibrated microphone-sound meter system. The 2 microphones will be suspended at a distance of 1 m approximately above the surface of the patient's bed. This arrangement allows a non-invasive measurement of snoring that simulates the distance between sleeping bed partners. Before every study the system would be acoustically calibrated using a reference noise produced by a noise generator (86 dB). The signal would be sent at a sampling rate of 12 KHz through an analogue-digital converter to a computer system for subsequent analysis. All digitized signals will be recorded in the hard disk of a personal computer. A noise analyzer (Praat; Boersma 2005) will be used for the intensity analysis of snoring sound (Boersma, 2005).

ELIGIBILITY:
Inclusion Criteria:

1. every night snoring;
2. no medication known to influence nasal resistance (e.g., antihistamines, vasoconstrictors, topical or systemic steroids);
3. no smoking for the last 6 months;
4. no upper or lower respiratory tract disease (e.g., upper respiratory tract infection, rhinitis, sinusitis, chronic obstructive pulmonary disease), including a history of nasal allergy; and
5. written informed consent from each patient.

Exclusion Criteria:

1. duration of snoring less than 60 minutes during sleep study, and
2. central apnoeas more than five percent of total apnoeas.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
snoring intensity | one week therapy
  Snoring intensity would be measured using a calibrated microphone-sound meter system

SECONDARY OUTCOMES:
snoring frequency | one week therapy
  Before and after each treatment regimen patients will undergo an assessment, which will consist of anterior rhinomanometry and polysomnography with concomitant measurement of snoring indices and breathing route pattern.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Koutsourelakis, MD, Principal Investigator — University of Athens
Locations (1):
- Department of Critical Care Medicine, Evangelismos Hospital of Athens, Athens, Greece

REFERENCES:
- [Background] Pevernagie D, Aarts RM, De Meyer M. The acoustics of snoring. Sleep Med Rev. 2010 Apr;14(2):131-44. doi: 10.1016/j.smrv.2009.06.002. Epub 2009 Aug 8. PMID 19665907